CLINICAL TRIAL: NCT02741388
Title: A Phase Ib Study of Oral Selinexor in Adult Patients With Relapsed/Refractory B-cell Lymphoma Receiving R-DHAOx or R-GDP
Acronym: SELINDA
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: The Lymphoma Academic Research Organisation (Other)
Collaborators: Karyopharm Therapeutics Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SELINDA
Record Dates: First submitted 2016-04-14; First posted 2016-04-18 (Estimated); Last update posted 2021-12-07 (Actual); Status verified 2021-12

CONDITIONS: B-cell Lymphoma
Keywords: selinexor; lymphoma; inhibitor of nuclear export
MeSH Terms: conditions — Lymphoma, B-Cell; Lymphoma | interventions — selinexor; Rituximab; Dexamethasone; Oxaliplatin; Cisplatin; Cytarabine; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Selinexor + immunochemotherapy (Experimental): Selinexor will be administered orally on Day1, 3, 8 and 10 of each 3-week cycle with an immunochemotherapy, R-DHAOx (Group A: rituximab + dexamethasone + oxaliplatin + cytarabine) or R-GDP (Group B: rituximab + dexamethasone + gemcitabine + cisplatin) for 3 cycles (choice of the immunochemotherapy left at the investigator's decision before patient's inclusion).
  Different dose levels of selinexor will be examined sequentially in each group: 20 mg flat (DL-1), 40 mg flat (DL1), 60 mg flat (DL2), 80 mg flat (DL3).
  Interventions: Drug: selinexor; Drug: Rituximab; Drug: Dexamethasone; Drug: Oxaliplatin; Drug: Cisplatin; Drug: Cytarabine; Drug: Gemcitabine

INTERVENTIONS:
Drug: selinexor
  Other Names: KPT-330
Drug: Rituximab
Drug: Dexamethasone
Drug: Oxaliplatin
Drug: Cisplatin
Drug: Cytarabine
Drug: Gemcitabine

SUMMARY:
This is an open label, multicenter, dose escalation, phase Ib study to determine the recommended phase II dose (RP2D), by assessing the maximum tolerated dose (MTD), safety and preliminary efficacy of selinexor in adult patients with relapsed/refractory B-cell malignancies receiving either R-DHAOx (Group A) or R-GDP (Group B). This dose escalation phase will be followed by an exploratory expansion phase in the same population with 12 patients enrolled in each group, who will receive selinexor at the RP2D.

The "3+3" design will be applied for dose escalation. The escalation will be performed independently in two distinct groups:

* Group A : Oral selinexor + R-DHAOx for 3 cycles (3-week cycles)
* Group B: Oral selinexor + R-GDP for 3 cycles (3-week cycles)

The choice of the conventional immunotherapy regimen which will be administered to each patient, R-DHAOx (Group A) or R-GDP (Group B), is left at the investigator's decision before patient's inclusion. Different dose levels for selinexor administration will be examined sequentially in each group by the Dose Escalation Committee (DEC): 4 doses of selinexor per 3-week cycle at 20 mg flat (Dose Level -1, DL-1), 40 mg flat (DL1), 60 mg flat (DL2) or 80 mg flat (DL3) will be taken orally by the patient on D1, D3, D8 and D10 of each cycle (dosing weeks = week 1 and week 2 of each 3-week cycle). Dose escalation will begin at DL1 and will continue until the MTD is exceeded or until the highest dose level defined in the study (DL3) is reached.

Dose escalation to the next planned dose level will be decided by the DEC based on the number of DLTs observed during the DLT assessment period.

The dose escalation phase will be followed by an exploratory expansion phase in the same two groups (Groups A and B), depending on the decision of the Independent Data Monitoring Committee (IDMC) after review of safety data at the end of dose escalation part.

Patients enrolled in the expansion phase will receive selinexor at the RP2D defined by the IDMC, together with either of the conventional regimen R-DHAOx or R-GDP (left at the investigator's choice).

ELIGIBILITY:
Inclusion Criteria:

1. Patients with any type of relapsed or refractory B-cell lymphoma
2. Eligible to receive R-DHAOx or R-GDP regarding the investigator's opinion
3. Who received prior therapy with at least one but no more than two lines therapies for B-Cell Lymphoma
4. Patient must have measurable disease defined by at least one single node or tumor lesion > 1.5 cm
5. Aged between 18 years and 70 years (included) on date of consent signature
6. Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1 or 2
7. With a life expectancy of ≥ 3 months
8. Having signed a written informed consent
9. Male patients (if sexually active with a woman of childbearing potential) must agree to use a reliable method of birth control during the study treatment and for at least 6 months after the last study drug administration. Male patients must agree to not donate sperm during the study treatment and for at least 6 months after the last study drug administration
10. Female patients of childbearing potential must agree to use two reliable methods of birth control during study treatment and for 6 months after the last dose and have a negative serum human chorionic gonadotropin (hCG) pregnancy test within 3 days prior to C1D1. Reliable methods of contraception include intrauterine devices, hormonal contraceptives [contraceptive pills, implants, transdermal patches, hormonal vaginal devices or injections with prolonged release], abstinence or sterilization of the partner.

Exclusion Criteria:

1. Previous treatment with selinexor
2. Known central nervous system or meningeal involvement by lymphoma
3. Contraindication to any drug contained in these regimen
4. Subjects with known Human Immunodeficiency Virus (HIV) positivity
5. Subjects with known active Hepatitis B (HB) infection (positive Ag HBs) or positive serology to hepatitis B (Ag HBs or antibody anti-HB c or positive DNA PCR) or active Hepatitis C (HCV) infection (patients with positive HCV serology are eligible only if PCR is negative for known HCV RNA)
6. Subjects with any uncontrolled active systemic infection requiring intravenous (IV) antibiotics
7. Any of the following laboratory abnormalities within 14 days prior to first administration (C1D1) of study treatment:

   1. Absolute neutrophil count (ANC) < 1,000 cells/mm3 (1.0 x 109/L)
   2. Spontaneous (within 7 days of any platelet transfusion) platelet count < 100,000/mm3 (100 x 109/L) (75 x 109/L if due to lymphoma)
   3. Aspartate aminotransferase (AST) or Alanine aminotransferase (ALT) > 5.0 x upper limit of normal (ULN)
   4. Serum total bilirubin > 2x Upper Limit of Normal (ULN), or > 5x ULN if due to Gilbert syndrome or lymphoma involvement
8. Creatinine clearance < 50 mL /min (for patients who will receive DHAOx) or < 70 mL/min (for GDP)
9. Subjects with pre-existing ≥ Grade 2 neuropathy
10. Prior history of malignancies other than lymphoma (except for basal cell or squamous cell carcinoma of the skin or in situ carcinoma of the cervix or breast) unless the subject has been free of the disease for ≥ 3 years
11. Any life-threatening illness, serious active disease or co-morbid medical condition, laboratory abnormality, organ system dysfunction or psychiatric illness which, in the investigator's opinion, could compromise the patient's safety, interfere with the absorption or metabolism of selinexor, or put the study outcomes at undue risk, or that would prevent the subject from signing the informed consent form
12. Pregnant or breastfeeding women
13. Use of any standard or experimental anti-cancer drug therapy within 28 days of the initiation (Day 1) of study drug therapy (administration of glucocorticoids should not exceed 1mg/kg/day in the 14 days prior to C1D1)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2021-09-29 (Actual); Study Completion 2021-09-29 (Actual)

PRIMARY OUTCOMES:
Incidence rate of dose-limiting toxicities (DLTs) observed during the DLT assessment period (cycle 1) at each dose level examined | Up to 35 days

SECONDARY OUTCOMES:
Response rates | 3 months
  Response rates will be evaluated according to the Lugano 2014 response criteria based on disease response assessment on Positron emission tomography-computed tomography (PET-CT) performed after completion of the 3 cycles of treatment (for patients who received all 3 cycles) or at permanent discontinuation of treatment (PTD evaluation, within 4 weeks after the last drug administration).
Duration of response | 3 years
  Duration of response is defined as the time of attainment of complete response (CR) or partial response (PR) to the date of first documented disease progression, relapse or death from any cause.
Progression-free survival (PFS) | 3 years
  PFS is defined as the time from inclusion into the study to the first observation of documented disease progression or death due to any cause.
Time to next anti-lymphoma treatment (TTNLT) | 3 years
  TTNLT is defined as the time from the date of inclusion to the date of first documented administration of any new anti-lymphoma treatment (chemotherapy, radiotherapy, radio-immunotherapy or immunotherapy, with the exception of High Dose Therapy/ASCT).
Overall survival (OS) | 3 years
  Overall survival is defined as the time from the date of inclusion to the date of death from any cause.
Incidence of grade ≥ 2 renal toxicities, grade ≥ 2 neuropathy, and grade ≥ 3 toxicities | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Hervé TILLY, MD, Study Chair — Centre Henri Becquerel, Rouen, France - LYSA; Marie MAEREVOET, MD, Study Chair — Institut Jules Bordet, Bruxelles, Belgium - LYSA
Locations (8):
- Institut Jules Bordet, Brussels, Belgium
- France (7):
  - CHU Dijon, Dijon
  - CHRU de Lille - Hôpital Claude Huriez, Lille
  - CHU Montpellier - Hôpital Saint Eloi, Montpellier
  - CHU Nancy - Hôpital de Brabois, Nancy
  - Hôpital Saint-Louis, Paris
  - CHU Bordeaux - Centre François Magendie, Pessac
  - Centre Henri Becquerel, Rouen

IPD SHARING:
Plan to Share IPD: No